CLINICAL TRIAL: NCT05275101
Title: Neural Mechanisms and Predictors of an Ultra-Brief Suicide Prevention Strategy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Stephanie M Gorka, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021H0039
Record Dates: First submitted 2022-02-10; First posted 2022-03-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Suicide
Keywords: Suicide Prevention; Crisis Response Planning; Suicide; functional magnetic resonance imaging
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Individuals who have not experienced suicidal ideation will not complete a suicide intervention.
- Crisis Response Planning (CRP) (Experimental): The crisis response planning (CRP) session will last between 30 minutes to 1-hour. It will occur face-to-face with a trained study therapist. The CRP session involves the following standard suicide intervention strategies: supportive listening, provision of crisis resources, and referral to a mental health professional (if not already established). The CRP active component involves a collaborative process in which the therapist invites the patient to share the events, symptoms, and contextual factors leading up to and surrounding the participant's suicidal crisis. Next, the patient and therapist identify the patient's personal warning signs for an emotional crisis, self-management coping skills, patient's reasons for living, and sources of social support. These components are written, by the patient, on an index card. The index card serves as a concrete reference for patients in the real-world.
  Interventions: Behavioral: Crisis Response Planning
- Crisis Risk Counseling (Active Comparator): The crisis risk counseling session will last between 30 minutes to 1-hour. It will occur face-to-face with a trained study therapist. It will include the following standard suicide intervention strategies: supportive listening, provision of crisis resources, and referral to a mental health professional (if not already established). The therapist will conduct a semi-structured suicide risk assessment interview, after which subjects will complete a self-guided safety plan worksheet. The worksheet takes approximately 10-minutes to complete and will be done independently.
  Interventions: Behavioral: Crisis Risk Counseling

INTERVENTIONS:
Behavioral: Crisis Response Planning — Individuals complete an experimental collaborative suicide intervention.
  Arms: Crisis Response Planning (CRP)
Behavioral: Crisis Risk Counseling — Individuals complete a standard crisis risk management intervention.
  Arms: Crisis Risk Counseling

SUMMARY:
The current study is a clinical trial, meaning a research study in which human subjects are prospectively assigned to one or more interventions to evaluate the effects of those interventions on health-related behavioral outcomes. Specifically, male and female adults with current suicidal intent will be randomly assigned to receive either a 1-hour session of crisis response planning (CRP) or a 1-hour session of standard crisis risk management (Treatment as Usual). The effects of both conditions on changes in emotion regulation, behavioral inhibition, stress reactivity, and suicide risk will be evaluated post-intervention and at six-month follow-up. Additional assessments of changes in mood and suicidality will be collected daily during the first 10-days following intervention, and then monthly for a duration of six months. A cohort of healthy controls is included in the study but are not randomized to either treatment condition. The investigators hypothesize the following: 1) A single session of CRP will acutely change suicide risk and 2) Individuals who receive CRP will show sustained improvements in measures of suicidality when compared to individuals who received the Treatment as Usual intervention.

ELIGIBILITY:
Inclusion Criteria:

* Generally medically and neurologically healthy
* Age 18 years or older at the time of consent
* Willing and able to give informed consent
* Individuals in the acutely suicidal group: endorse current suicide intent as indicated by a total score of 5 or greater on the Beck's Scale for Suicidal Ideation.

Exclusion Criteria:

* Medical or neurologic condition or neurocognitive dysfunction that would interfere with the study
* Current or past manic/hypomanic episode, schizophrenia, or psychotic symptoms
* Deafness in either ear
* Currently pregnant or trying to become pregnant
* Electroconvulsive therapy (ECT) within the past 6 months
* Current moderate to severe substance use disorder
* Lack of fluency in English
* Positive alcohol breathalyzer test and/or acute drug intoxication the day of the fMRI scans
* Unwilling or unable to sign the informed consent document
* Under 18 years old at the time of enrollment
* Traumatic brain injury from a suicide attempt or another event
* Presence of ferrous-containing metals within the body
* Inability to tolerate small, enclosed spaces without significant anxiety
* Individuals enrolled as controls: no lifetime history of any DSM-5 disorder
* Individuals enrolled as controls: no lifetime history of suicide ideation or intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Frontolimbic neural circuit activation and connectivity | Pre-treatment, Post-treatment, and 6-months follow-up.
  Task-induced activity in frontolimbic neural circuits measured with fMRI. Core regions of interest are: ventral prefrontal cortex, dorsal prefrontal cortex, inferior frontal gyrus, insula, and dorsal anterior cingulate cortex.
Suicidality | Pre-treatment, Post-treatment, 1-week post-intervention, monthly post-intervention, and 6-months post-intervention.
  Self-reported suicide ideation, intent, behaviors and urges will be repeatedly assessed throughout the protocol using the Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R), Beck's Scale for Suicidal Ideation (SSI), Lethality Rating Scale, and Suicide Cognitions Scale - Revised (SCS-R).

SECONDARY OUTCOMES:
Markers of negative affectivity | Pre-treatment, Post-treatment, and 6-months follow-up.
  Acoustic startle electromyographic (EMG) response, behavioral data (i.e., reaction times and self-report scales) during lab tasks.
Mood and psychiatric symptoms | Pre-treatment, Post-treatment, 1-week post-intervention, monthly post-intervention, and 6-months post-intervention.
  Mood states and general depression and anxiety symptoms are repeatedly assessed throughout the protocol using the Beck Depression Inventory (BDI-II), Beck Anxiety Inventory (BAI), Beck Hopelessness Scale, Snaith-Hamilton Pleasure Scale (SHAPS), UPPS-P Impulsive Behavior Scale, and Validated Visual Mood Analog Scales (VMAS).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gorka, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, including fMRI, startle eyeblink, and behavior, from this project will be submitted to the NIMH Data Archive (NDA) at the subject level along with appropriate supporting documentation to enable efficient use of the data by the research community. We will follow instructions as discussed in the NIMH Data Archive Data Sharing Terms and Conditions.
  We will follow the two-tier procedure described in the guidelines:
  1. Raw continuous fMRI recordings will be submitted in standard formats (Matlab mat format, DICOM format and NIFTI format). Experimental condition information will be supplied in text format along with other critical information.
  2. Analyzed data (BOLD data, BOLD-startle eyeblink data) associated with a manuscript will be shared as soon as possible, and at the latest, at the time of publication of the manuscript. These data may be accompanied, if applicable, by other data such as behavioral data, supplied in text format.
Time Frame: The data, as outlined above, will be submitted to the NIMH Data Archive biannually per NIMH requirements throughout the duration of the study.
URL: https://nda.nih.gov/